CLINICAL TRIAL: NCT04770571
Title: A Prospective, Multicenter Study Evaluating the Safety and Performance of Posterior Fixation in Trauma, Reconstructive, and Tumor Surgery of the Occipito-cervico-thoracic Spine
Brief Title: Posterior Cervical Fixation Study
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.PCF1020
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Craniocervical Injuries; Cervical Radiculopathy; Cervical Disc Disease; Cervical Fusion; Cervical Spine Disease; Cervical Myelopathy; Cervical Instabilities Spine; Thoracic Injury
MeSH Terms: conditions — Intervertebral Disc Degeneration; Trauma, Nervous System; Radiculopathy; Klippel-Feil Syndrome; Thoracic Injuries | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Vuepoint II OCT
  Interventions: Device: observational study
- Reline-C
  Interventions: Device: observational study

INTERVENTIONS:
Device: observational study — observational

SUMMARY:
The objective of this study is to evaluate the safety and performance of occipito-cervico-thoracic spine surgery using posterior fixation as measured by reported complications, radiographic outcomes, and patients reported outcomes (PROs).This study is being undertaken to identify possible residual risks and to clarify mid-to long-term clinical performance that may affect the benefit/risk ratio of posterior fixation systems.

DETAILED DESCRIPTION:
This study is a prospective, uncontrolled, multicenter study to evaluate the safety and performance of select occipito-cervico-thoracic posterior fixation systems in patients who undergo posterior fixation fusion surgery. Consecutive patients at a given site who meet eligibility requirements will be asked to consent to participate in the study. These patients will present with traumatic, reconstructive, and/or tumor conditions in the craniocervical, cervical, and/or upper thoracic spine that are amenable to surgical treatment and will be screened prior to study enrollment. Once enrolled in the study, subjects will undergo posterior occipito-cervico-thoracic fixation surgery using one of the NuVasive posterior fixation systems (Vuepoint II OCT or Reline-C) based on the surgeon's standard of care. At least 150 subjects (a minimum of 75 in each implant arm) will be enrolled and will be followed for 24 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥18 years of age at the time of consent
2. Have planned craniocervical, cervical (C1 to C7), and/or upper thoracic (T1-T3) spine surgery using posterior fixation planned for treatment of any of the following conditions:

   1. traumatic spinal fractures and/or traumatic dislocations
   2. instability or deformity
   3. failed previous fusions (e.g., pseudoarthrosis)
   4. tumors involving the cervical spine
   5. degenerative disease, including intractable radiculopathy and/or myelopathy, neck and/or arm pain of discogenic origin as confirmed by radiographic studies, and degenerative disease of the facets with instability
3. Using one of the following posterior occipito-cervico-thoracic fixation systems (NuVasive, Inc, San Diego, CA):

   1. Vuepoint II OCT
   2. Reline-C
4. Able to undergo surgery based on physical exam, medical history, and surgeon judgment
5. Understands the conditions of enrollment and is willing to sign an informed consent form to participate in the study

Exclusion Criteria:

1. Patient is involved in active litigation relating to the spine (workers' compensation claim is allowed if it is not contested)
2. Use of bone growth stimulators postoperatively
3. Active smoking within 6 weeks of surgery
4. Patient has known sensitivity to materials implanted
5. Systemic or local infection (latent or active) or signs of local inflammation
6. Patient has inadequate bone stock or quality, or a physical or medical condition that would prohibit beneficial surgical outcome based on surgeon judgment
7. Pregnant, or plans to become pregnant
8. Patient is a prisoner
9. Patient is participating in another clinical study that would confound study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled Population
  The Enrolled Population will include all subjects who meet the criteria for enrollment, specifically, those subjects who:
  * Satisfied the inclusion and exclusion criteria,
  * Signed the informed consent, and
  * Underwent the surgical procedure, as defined in this protocol.
  Evaluable Population
  The Evaluable Populations will include all subjects who:
  * Were included in the Enrolled Populations,
  * Completed the study, and
  * Had no major protocol deviations.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Complications of Posterior Fixation System | 24 months
  Rate of complications (i.e., safety) attributable to the use of the associated posterior fixation system.
Radiographic Success | 24 months
  The proportion of subjects with apparent radiographic success at:
  1. Latest timepoint available for patients undergoing surgery to treat advanced stage tumors
  2. 24 months postoperative for subjects undergoing surgery to treat instabilities, traumatic spinal fractures, failed previous fusions, or degenerative disease

SECONDARY OUTCOMES:
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for neck/arm pain measured by visual analog scale (VAS). | 24 months
  Neck and arm pain measured using a visual analog scale (VAS) will be assessed to determine the percentage of subjects who meet MCID (2.5 points and 2.5 points respectively) where 0 is "No Pain" and 10 is "Unbearable Pain".
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for disability measured by the neck disability index. | 24 months
  Disability measured by the neck disability index (NDI) will be assessed to determine the percentage of subjects who meet MCID (7.5 points) where a higher score on the NDI indicates a more severe disability.
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline measured by overall physical and mental health from PROMIS-10. | 24 months
  Overall physical and mental health measured by PROMIS-10 will be assessed to determine the percentage of subjects who meet MCID (5 points). PROMIS-10 scoring uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
Percentage of subjects meeting substantial clinical benefit (SCB) for neck/arm pain as compared to baseline for neck/arm pain measured by visual analog scale (VAS). | 24 months
  Neck and arm pain measured using a visual analog scale (VAS) will be assessed to determine the percentage of subjects who meet SCB (3.5 points) where 0 is "No Pain" and 10 is "Unbearable Pain".
Percentage of subjects meeting substantial clinical benefit (SCB) as compared to baseline for disability measured by the neck disability index. | 24 months
  Disability measured by the neck disability index (NDI) will be assessed to determine the percentage of subjects who meet SCB (9.5 points) where a higher score on the NDI indicates a more severe disability.
Percentage of subjects meeting substantial clinical benefit (SCB) as compared to baseline measured by overall physical and mental health from PROMIS-10. | 24 months
  Overall physical and mental health measured by PROMIS-10 will be assessed to determine the percentage of subjects who meet SCB (6.8 points). PROMIS-10 scoring uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
Rate of complications attributable to the use of any additional NuVasive instruments, implants, or technologies | 24 months
  Rate of complications attributable to the use of any additional NuVasive instruments, implants, or technologies.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — NuVasive
Locations (7):
- United States (7):
  - UC Irvine Medical Center, Orange, California
  - Hartford Healthcare Bone & Joint Institute, Hartford, Connecticut
  - MedStar Health Research Institute, Hyattsville, Maryland
  - NY Spine Institute, New York, New York
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No